CLINICAL TRIAL: NCT02189057
Title: A Pharmacokinetic/Pharmacodynamic Genetic Variation Treatment Algorithm Versus Treatment As Usual for Management of Depression
Acronym: MOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Frye, Chair-Psychiatry/Psychology, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-007981
Record Dates: First submitted 2014-07-08; First posted 2014-07-14 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Depression; Mood Disorder; Bipolar
Keywords: Bipolar; Unipolar; Genotyping; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Depression; Mood Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either genotyping intervention or treatment as usual.
Who Masked: Participant, Investigator
Masking Description: Subject and study staff will be blind to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GeneSight guided treatment (Experimental): GeneSight guided group will have their research psychiatrist make treatment recommendations based on AssureRx GeneSight genotyping results.
  Interventions: Other: AssureRx GeneSight genotyping results
- Treatment as usual group (Active Comparator): Treatment as usual group will have treatment recommendations based on clinical judgment
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: AssureRx GeneSight genotyping results
  Arms: GeneSight guided treatment
Other: Treatment as usual
  Arms: Treatment as usual group

SUMMARY:
The overall goal of this investigator-initiated trial is to evaluate the treatment outcome of depression utilizing platform algorithm products that can allow rapid identification of pharmacokinetic (PK) and/or pharmacodynamic (PD) genomic variation. This new technology may have the potential to optimize treatment selection by improving response, minimizing unfavorable adverse events / side effects and increasing treatment adherence.

DETAILED DESCRIPTION:
Treatment seeking depressed patients (SCID confirmed major depressive disorder or bipolar I/II disorder) to the Mayo Clinic Depression Center will be invited to participate in this study evaluating the Assurex GeneSight® platform; this new technology can rapidly assess PK and PD genetic variation that can potentially impact antidepressant, antipsychotic, and stimulant associated treatment outcomes for depression. This study will recruit treatment seeking patients with major depression with an index episode of moderate symptom severity that has been unresponsive or poorly tolerated to at least one prior antidepressant treatment. This will be an 8-week, double-blind trial where depressed patients are randomized to testing results of GeneSight® (tricolored clinical report) prior to treatment selection (n=138) vs. treatment as usual (tricolored dummy report) (n=138). All testing results will be made available after the 8-week trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, male or female, any race/ethnicity
2. Mayo Clinic Depression Center inpatient or outpatient, or an outpatient of Mayo Clinic Rochester and satellite clinics, and outpatients from Mayo Clinic Health System clinics
3. Ability to provide informed consent
4. Structured Clinical Interview (SCID) confirmed major depressive episode associated with Major Depressive Disorder, Bipolar I/II disorder, or Schizoaffective Bipolar Disorder
5. Current index episode of major depression < 2 years duration
6. Moderate symptom severity defined by HAMD-17 rating scale score ≥ 17 [8]
7. Current index episode having not been treated with psychotropic medications or inadequately responsive to treatment (IRT). IRT defined as intolerability, adverse event, or inadequate efficacy of current psychotropic medication (at least 4 weeks duration)
8. Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study, including all visits and tests
9. Negative serum or urine pregnancy test (or history of hysterectomy)
10. Negative urine toxicology test (will only be completed at the request of the treating clinician).

Exclusion Criteria:

1. Inability to speak English
2. Inability or lack of willingness to provide informed consent
3. Axis I or II disorder other than depression (i.e., by clinical assessment) that is the primary reason for treatment
4. Psychotropic medication change (including dosage) between screening & baseline visit with exception of no more than 8mg of Ativan within a 24-hour period.
5. Patients who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria for any significant current substance use disorder other than nicotine or caffeine. Must have at least early, partial or full, remission X 3 months
6. Clinically diagnosed cannabis use disorder, or SCID confirmed cannabis abuse or dependence.
7. Current clinical diagnosis delirium, dementia, other cognitive disorders, or non-mood psychotic disorder (i.e., schizophrenia, delusional disorder)
8. Index episode symptoms of hallucinations or delusions
9. Serious suicidal risk and/or in need of immediate hospitalization as judged by the investigator
10. History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 6 months
11. Significant unstable medical condition
12. Hepatic insufficiency (2.5 X upper limit of normal (ULN) for Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ), past liver transplant recipient, and/or clinical diagnosis of cirrhosis of the liver
13. Malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening; malignancy more than 1 year prior to screening must have been local and without metastasis and/or recurrence, and if treated with chemotherapy, without nervous system complications
14. Participation in another clinical trial within 30 days of the screening visit
15. Anticipated inability to attend scheduled study visits
16. Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol
17. Known cytochrome (CYP) & serotonin transporter genomic testing results within 5 years
18. A score of ≥15 on the Young Mania Rating Scale (YMRS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Change in depression as measured by the Quick Inventory of Depressive Symptoms (QIDS-C16) | baseline, 8 weeks
  The QIDS-C16 is a 16-item scale that is clinician-rated; it is designed to assess the severity of depressive symptoms. The QIDS-C16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression. A negative change indicates improvement in the subject's depression, and a positive change indicates a worsening of the subject's depression.

SECONDARY OUTCOMES:
Number of subjects with improvement of depressive symptoms as shown by 50% reduction in QIDS-C16 score | 8 weeks
  The QIDS-C16 is a 16-item scale that is clinician-rated; it is designed to assess the severity of depressive symptoms. The QIDS-C16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression. A negative change indicates improvement in the subject's depression, and a positive change indicates a worsening of the subject's depression.
Number of subjects with improvement of depressive symptoms as shown by a score <6 on QIDS-C16 | 8 weeks
  The QIDS-C16 is a 16-item scale that is clinician-rated; it is designed to assess the severity of depressive symptoms. The QIDS-C16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression. A negative change indicates improvement in the subject's depression, and a positive change indicates a worsening of the subject's depression.
Number of subjects with improvement of depressive symptoms as shown by score of "much" or "very much improved" on Clinical Global Impression - Improvement Scale | 8 weeks
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1. Very much improved, 2. Much improved, 3. Minimally improved, 4. No change, 5. Minimally worse, 6. Much worse, 7. Very much worse
Improvement of depressive symptoms as shown by the Hamilton Rating Scale for Depression (HAMD-17) | 8 weeks
  The HAMD-17 is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. The 17 items are rated on either a 5-point (0-4) or a 3-point (0-2) scale. In general, the 5 point scale items use a rating of 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. The 3-point scale items use a rating of 0=absent; 1=probable or mild; 2=definite. The total HAMD-17 score ranges from 0 (not ill) to 52 (severely ill). A negative change indicates improvement in the subject's depression/anxiety symptoms, and a positive change indicates a worsening of the subject's depression/anxiety symptoms.
Improvement of depressive symptoms | 8 weeks
  Treatment adherence based on concordance vs. non-concordance of gene test results and clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States